CLINICAL TRIAL: NCT05333692
Title: Oral Nutritional Supplementation of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi Taiwan Ltd. (Industry)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FrPE-005-IEN
Record Dates: First submitted 2022-04-07; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEPRO® (Active Comparator)
  Interventions: Dietary Supplement: NEPRO® , Abbott
- Fresubin® Protein Energy DRINK (Experimental)
  Interventions: Dietary Supplement: Fresubin® Protein Energy DRINK

INTERVENTIONS:
Dietary Supplement: Fresubin® Protein Energy DRINK — 1-2 bottles of Fresubin® Protein Energy DRINK per day
  Arms: Fresubin® Protein Energy DRINK
Dietary Supplement: NEPRO® , Abbott — 2-4 cans NEPRO® per day
  Arms: NEPRO®

SUMMARY:
This study is aimed to demonstrate that increase in serum albumin concentration (week 8 -baseline) after test treatment (Fresubin® Protein Energy DRINK), a standard ONS, is not relevantly smaller than that after control treatment with NEPRO®.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years
2. Acute or chronic renal failure patients who need dialysis and already dialysis for 3 months at least.
3. Malnutrition patients. Definition of Malnutrition is serum albumin level<3.5g/dL, calorie digestion below 35kcal/IBW or protein digestion below 1.2g/IBW.

Exclusion Criteria:

1. BMI<18.5 and calorie intake unable to reach 50% of the recommended level
2. BMI>30 kg/m2,
3. abnormal liver function,
4. malignant disease,
5. scheduled surgery within a month or after surgery,
6. infectious disease,
7. suboptimal tolerance of nutritional supplements,
8. inflammatory bowel disease, bowel obstruction,
9. acute condition complicated with multiple organ failure or under palliative care.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Serum Albumin level change | baseline, weerk 4 and week 8

SECONDARY OUTCOMES:
Body Weight (kg) and Height(cm) change, and these results will be combine to report BMI (kg/m^2) change | baseline, weerk 4 and week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No